CLINICAL TRIAL: NCT00040482
Title: Intensive Immunosuppression Followed by Rescue With CD34 Selected, T Cell Depleted, Leukopheresis Products in Patients With Multiple Sclerosis
Brief Title: High Dose Chemo/Radiotherapy and Hematopoietic Stem Cell Transplant for Patients With Multiple Sclerosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: The Methodist Hospital Research Institute (Other); Center for Cell and Gene Therapy, Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Robert Krance, Professor, Pediatrics-Hem-Onc Cell & Gene, Baylor College of Medicine
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H7156; Multiple Sclerosis
Record Dates: First submitted 2002-06-26; First posted 2002-06-28 (Estimated); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — Cyclophosphamide; Mesna; Radiotherapy

INTERVENTIONS:
Drug: Cyclophosphamide
Drug: ATG
Drug: MESNA
Procedure: Radiation therapy

SUMMARY:
Multiple Sclerosis is a disease that may be caused by the immune system reacting against the nervous system. It is possible, that by changing the immune system we can modify the progression of this disease. In this study, we will try to learn whether treatment with a bone marrow transplant (BMT) can help patients with multiple sclerosis. We will also try to learn what the side effects are of this treatment in patients with multiple sclerosis.

DETAILED DESCRIPTION:
To participate in this study, patients will need to have a central line (a thin plastic catheter or tube that is placed during surgery into one of the large veins in the neck or chest). Central lines are used to give intravenous medications or to draw blood. Before the transplant we will test the patients blood for viruses which can cause problems after the transplant. These viruses include Hepatitis B, which causes liver damage, cytomegalovirus, which causes lung disease and HIV which causes AIDS. If a patient is positive for the AIDS virus, they will not be able to undertake the transplant. In addition to these blood tests patients will also have an MRI (where pictures are created using magnetic rather than x-ray energy) of the brain and other evaluations that are standard for any patient before having a transplant.

Before the transplant patients will receive daily G-CSF (Neupogen). This medicine will help to stimulate the production of white blood cells (WBC) that will be used for the bone marrow transplant. In addition, 6 tablespoons of blood will be collected to look at how the immune system is functioning before and after transplant. After the white blood cells have reached a certain level, patients will undergo leukapheresis. Leukapheresis is a procedure where blood is removed from a patients arm, pumped into a machine where the white blood cells are separated from most of the other cells, then returned to the patient through the same needle or through a needle in the other arm. After collection of the white blood cells, we will use a device in the lab to select out certain types of white blood cells (CD34+).

After leukapheresis, patients will receive an antibody from horses called Atgam (ATG) to help destroy the immune system and also a drug called cyclophosphamide. After this, radiation treatment will be given to the entire body. This will be done 2 times a day for 3 days. This treatment will kill most of the blood-forming cells in the bone marrow. We will then give the CD34+ white blood cells that were collected during leukapheresis.

Blood will be collected for immune reconstitution studies monthly for 3 months and at 6, 9, and 12 months after transplant to look at how the immune system is functioning. The amount of blood taken will be no more than 90ml (6 tablespoons). After the first year of treatment patients will continue to have 90ml (6 tablespoons) of blood taken for immune reconstitution studies every 6 months for 2 more years.

ELIGIBILITY:
Inclusion:

* The diagnosis of primary or secondary progressive multiple sclerosis or relapsing-remitting multiple sclerosis. Patients with relapsing/remitting MS should demonstrate sustained accumulated disability based upon accepted standard. Relapsing/remitting MS is characterized by unpredictable recurrent attacks of neurologic dysfunction followed by complete, partial or no recovery.
* By the Expanded Disability Status Scale (EDSS) the measure of disability equals or exceeds 5.0 but does not exceed 7.5.
* For primary or secondary progressive MS, the progression of disease using EDSS criteria during the proceeding 12 months equals or exceeds 1.0.
* Symptoms and manifestations of MS activity have not responded to conventional treatment, e.g. high dose prednisone, beta interferon, conventional dose cytoxan, glatiramer acetate etc.
* The patient is able to undergo collection of sufficient numbers of HSCs to meet protocol requirements, i.e. 3X10e6 CD34+ cells.
* Males and females <60 years old.
* Patient must have a life expectance of >6 weeks.
* Patients should not have received prior lymphoid irradiation.
* Patients should not have a history of hypersensitivity to murine proteins or E.coli derived proteins.
* Patients should not have a history of lack of compliance with medical care or any medical or psychiatric conditions which would compromise their ability to comply with the protocol.
* Patients should not have evidence of myelodysplasia or an active malignancy.
* Patients should not be receiving concurrent beta interferon therapy or high dose prednisone.
* The patient does not exhibit significant organ toxicity from any cause. Significant organ toxicity includes:- Creatinine greater than twice normal; glomerular filtration rate less than 40 ml/min. - FEV1 or FVC less than 75% predicted; DLCO less than 50% predicted.- Significant cardiac dysfunction defined as life endangering arrythmias or a shortened ejection fraction(less than 26%).- Hepatic transaminases greater than two times normal; total bilirubin greater than 3.0 mg/dl.
* The patients are able to give informed consent.
* Both male and female patients must agree to use effective contraception for a minimum of 12 months post transplant. Effective contraception includes total abstinence, oral contraceptives, an intrauterine device, contraceptive implants under the skin (Norplants), contraceptive injections, or contraceptive foam with a condom. In addition, the male partner should use a condom.

Exclusion:

* Active infection.
* Unable to tolerate an MRI.
* HIV positive patient.
* Pregnant and lactating women

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10
Dates: Start 1999-04; Study Completion 2005-08

CONTACTS AND LOCATIONS:
Overall Officials: Malcolm K. Brenner, MD, Study Chair — Baylor College of Medicine
Locations (1):
- The Methodist Hospital, Houston, Texas, United States